CLINICAL TRIAL: NCT00553839
Title: Pharmacokinetics of Ketamine in Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Chandra Ramamoorthy, Professor of Anesthesia, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3384; NCT01100138 (obsolete NCT alias)
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2014-08

CONDITIONS: The Pk of IV Ketamine in Children With Heart Disease
Keywords: anesthesia; children; ketamine; pharmacokinetics
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine (Other): Then a 2 mg/kg IV bolus of Ketamine hydrochloride will be given as part of general anesthesia for procedure
  Interventions: Drug: ketamine hydrochloride

INTERVENTIONS:
Drug: ketamine hydrochloride — Open label pharmacokinetic study to be conducted in infants and children presenting for medical procedures (eg., surgery or cardiac catheterization). After the start of the procedure, a 0.5 cc preload blood sample (T0) will be drawn from an IV line. Then a 2 mg/kg IV bolus of Ketamine will be administered over 5 minutes. Timed 0.5 ml blood samples will be drawn at the following intervals: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus.

SUMMARY:
Dosing of medications is based on the plasma level achieved with a given dose and how long the medicine remains in the body. This study is called pharmacokinetics-that is, what the body does to the medication. Ketamine is an intravenous medication used for anesthesia and sedation in children. However the pharmacokinetics of Ketamine has not been systematically studied. We propose to study the pharmacokinetics of ketamine in different age groups of children ranging from infants to teenagers.

DETAILED DESCRIPTION:
This is an open label study that will be conducted in infants and children presenting for procedures (eg., surgery or cardiac catheterization) at Stanford and Lucile Packard Children's hospital in California and at The Children's Hospital in Denver, CO. Patients with abnormal kidney or liver functions will be excluded from the study as the dysfunction in these organs affects the clearance of medications from the body and affects dosing. Preterm neonates will also be excluded. All patients will be premedicated and anesthetised at the discretion of the anesthesia faculty providing clinical care for the child. Once the patient's procedure is underway, a 0.5 cc blood sample will be drawn from an intravenous line. This is the preload blood sample (T0). Following this a 2mg/kg intravenous bolus of Ketamine will be administered over 5 minutes (this is the usual dose and manner in which ketamine is administered). Five minutes after the bolus, timed blood samples will be drawn at the following intervals: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus. (Total 14 blood samples; total blood required is 7 mls for the entire study). When the procedure is completed the anesthesiologist will awaken the patient as per their usual practice. Blood samples that still need drawing will be done in the post-anesthesia recovery room or intensive care or ward-any location where the patient is likely to remain after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (38 weeks gestation)and infants and children up to age 18 years.
* Patients who require procedures that necessitate at least 8 hours in the hospital and those being admitted after procedure will be eligible to participate.
* Patients who will receive ketamine as part of their standard anesthesia regimen.

Exclusion Criteria:

* Preterm neonates
* Liver Disease
* Kidney disease
* Heart failure
* Sepsis
* Patients receiving anticonvulsants or barbiturates

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Ramamoorthy, MBBS, FRCA, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital, Denver, Colorado

REFERENCES:
- [Result] Elkomy MH, Drover DR, Hammer GB, Galinkin JL, Ramamoorthy C. Population pharmacokinetics of ketamine in children with heart disease. Int J Pharm. 2015 Jan 15;478(1):223-231. doi: 10.1016/j.ijpharm.2014.11.026. Epub 2014 Nov 13. PMID 25448584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group Assignment
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children between 6 months to 18 years of age with cardiac diseases in order to rationalize an effective 2-h anesthetic medication personalized based on cardiac function and age
Groups:
- Ketamine: Then a 2 mg/kg IV bolus of Ketamine hydrochloride will be given.
  ketamine hydrochloride: Open label pharmacokinetic study to be conducted in infants and children presenting for medical procedures (eg., surgery or cardiac catheterization). After the start of the procedure, a 0.5 cc preload blood sample (T0) will be drawn from an IV line. Then a 2 mg/kg IV bolus of Ketamine will be administered over 5 minutes. Timed 0.5 ml blood samples will be drawn at the following intervals: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus.
Arm/Group | Ketamine
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.44 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Clearance and Intercompartmental Clearance
Description: pK analysis of ketamine in children with pre-existing congenital heart disease following a single dose of ketamine in order to rationalize an effective 2-h anesthetic medication, personalized based on cardiac function and age.
  Total Clearance and Intercompartmental Clearance were analyzed using Bootstrap model.
Time Frame: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus.
Population: Children up to 18 years of age children with pre-existing congenital heart disease
Measure: Median (95% Confidence Interval); unit: L/h/70kg
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 21
L/h/70kg
  Total Clearance | 60.0 [51.4 to 72.0]
  Intercompartmental Clearance | 70.8 [49.7 to 106]

2. Primary Outcome: Central and Peripheral Volume of Distribution
Description: pK analysis of ketamine in children with pre-existing congenital heart disease following a single dose of ketamine in order to rationalize an effective 2-h anesthetic medication, personalized based on cardiac function and age.
  Central and Peripheral Volume of Distribution were analyzed using Bootstrap model.
Time Frame: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus.
Population: Children up to 18 years of age children with pre-existing congenital heart disease
Measure: Median (95% Confidence Interval); unit: L/70kg
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 21
L/70kg
  Central Volume of Distribution | 57.6 [45.0 to 82.6]
  Peripheral Volume of Distribution | 149 [114 to 206]

3. Primary Outcome: Residual Error
Description: pK analysis of ketamine in children with pre-existing congenital heart disease following a single dose of ketamine in order to rationalize an effective 2-h anesthetic medication, personalized based on cardiac function and age.
  Residual Error was analyzed using Bootstrap model.
Time Frame: 5, 10, 15, 20, 30, 45, 60, 120, 180, 240, 300, 360 and 720 minutes after bolus.
Population: Children up to 18 years of age children with pre-existing congenital heart disease
Measure: Median (95% Confidence Interval); unit: proportional %
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 21
proportional % | 16.1 [13.4 to 18.7]

ADVERSE EVENTS:
Arm/Group | Single Group Assignment
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No